CLINICAL TRIAL: NCT00063713
Title: A Phase 2 Study of VELCADE in Subjects With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: VELCADE in Subjects With Relapsed or Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M34103-053; NCT00084851 (obsolete NCT alias)
Record Dates: First submitted 2003-07-02; First posted 2003-07-04 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib; WW Domain-Containing Oxidoreductase

INTERVENTIONS:
Drug: VELCADE TM (bortezomib) for Injection

SUMMARY:
The purpose of this study is to find out whether treatment with VELCADE will increase the time it takes for lymphoma to get worse.

DETAILED DESCRIPTION:
VELCADE is approved in multiple myeloma for patients who have received two prior therapies and their disease came back or got worse while on their second therapy. VELCADE is currently being studied in other types of cancers.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older
* Confirmed diagnosis of mantle cell lymphoma
* Documented relapse or progressive disease following 1 or 2 prior lines of anti-cancer therapy. At least one of those regimens must have included an anthracycline or mitoxantrone. Relapsed or progressive disease, since last therapy must be documented by new lesions or objective evidence of the progression of existing lesions.
* At least 1 measurable or evaluable site of disease
* Voluntary consent

Exclusion Criteria

* Previous treatment with VELCADE
* Any experimental or anti-cancer therapy within 3 weeks before the first dose of study drug
* Radiation therapy within 3 weeks before the first dose of study drug
* Major surgery with 2 weeks before the first dose of study drug
* Rituximab, Campath, or other unconjugated therapeutic antibody within 4 weeks before the first dose of study drug
* Radioimmunotherapy or other toxin immunoconjugates such as Zevalin or Bexxar within 10 weeks before the first dose of study drug
* History of allergic reactions to boron or mannitol compounds
* Diagnosed or treated for another malignancy other than mantle cell lymphoma with 5 years before the first dose of study drug
* Active systemic infection requiring treatment
* Women patients must not be pregnant or breast-feeding, confirmed through pregnancy test obtained during screening (this test is not required for women who are post-menopausal or surgically sterile)
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Concurrent treatment with another investigational drug or participation in non-treatment studies is not allowed if it interferes with participation in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152
Dates: Start 2003-06; Primary Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - University of Alabama, Birmingham, Alabama
  - Alta Bates Medical Center, Berkeley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda Cancer Research Institute, Loma Linda, California
  - UCLA School of Medicine, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado Cancer, Denver, Colorado
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - The Rush Cancer Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospital Division, Iowa City, Iowa
  - North Memorial Hospital, Robbinsdale, Minnesota
  - Onc/Hem Associates of Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Beth Israel Medical Center, New York, New York
  - St Lukes-Roosevelt Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Hospital Cornell Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest, University health Sciences/Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Oregon Health Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University Hospital-Madison Wisconsin, Madison, Wisconsin